CLINICAL TRIAL: NCT07003009
Title: Detection of Lymph Node Positivity in Patients With Invasive Ductal Breast Cancer Using Immun Checkpoint Washout
Brief Title: Immun Checkpoint Washout in Patients With Invasive Ductal Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Chief of General Surgery, Principal Investigator, Clinical Associate professor, Istanbul Training and Research Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Breast lymph node
Record Dates: First submitted 2025-03-03; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Metastatic; Breast Carcinoma
Keywords: Immune checkpoints; Breast Cancer; Lymph node; Washout
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Intervention Model Description: A washout sample will be obtained by axillary lymph nodes suspected to be metastatic which is not performed in routine lymph node biopsy procedure. Similarly, an axillary lymph node that is deemed non-metastatic based on imaging findings will be sampled under ultrasound guidance for the same patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metastatic axillary lymph nodes suspected (Experimental)
  Interventions: Diagnostic Test: Malign Lymph Node Washout
- Benign lymph nodes (Other)
  Interventions: Diagnostic Test: Benign Lymph Node Washout

INTERVENTIONS:
Diagnostic Test: Malign Lymph Node Washout — During routine axillary lymph node sampling, which is performed as part of standard staging using imaging methods, a washout sample (which is not not routinely applied ) will be obtained by injecting 1 cc of 0.9% saline into axillary lymph nodes suspected to be metastatic. The aspirated washout sample will be placed in a biochemistry gel tube labeled as Sample 1.
  Other Names: Fine needle aspiration biopsy; Washout
  Arms: Metastatic axillary lymph nodes suspected
Diagnostic Test: Benign Lymph Node Washout — Description: During the biopsy performed to histopathologically confirm the benign nature of a radiologically presumed benign axillary lymph node, a washout sampling will also be conducted by injecting 1 cc of 0.9% saline into benign lymph node. The aspirated washout sample will be placed in a biochemistry gel tube labeled as Sample 2.
  Other Names: Fine needle aspiration biopsy; Washout
  Arms: Benign lymph nodes

SUMMARY:
Invasive ductal carcinoma is the most common type of invasive breast cancer. In cases where axillary lymph node metastases are diagnosed through screening, they can be found in up to 25% of cases, and in symptomatic cases, up to 60% of cases. The clinical detection accuracy of axillary lymph node metastases is only 33%. Accurate staging of lymph nodes in breast cancer patients is crucial for both prognosis and treatment. Ultrasonography is much more sensitive than physical examination alone for determining axillary lymph node involvement in breast cancer staging. Fine needle aspiration biopsy or core biopsy is diagnostic in lymph nodes that cannot be clarified solely by ultrasonography or are suspicious. Although biopsy sampling yields high diagnostic rates, it requires an experienced pathologist and sometimes takes weeks to yield results. Therefore, there is a need for faster and less costly diagnostic methods for diagnosing axillary metastases. Among thyroid cancers, papillary thyroid carcinomas, a malignancy in which the lymph node washout method is used to determine lymph node metastasis, are the most common. In papillary thyroid cancer patients, washout sampling of neck lymph nodes by fine needle aspiration, searching for thyroglobulin, a protein normally found in thyroid tissue, is considered one of the most valid methods for detecting lymph node metastasis in this cancer. In recent years, immune checkpoint molecules associated with cancer have been widely used as biomarkers and agents in both diagnosis and treatment for cancer patients. There are numerous publications in the literature regarding the expression of immune checkpoint molecules such as Programmed cell death protein 1 (PD-1), Programmed death ligand 1 (PD-L1), and The cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) on the cell surface of breast cancer patients. Although the natural soluble forms of receptors and ligands of immune checkpoint molecules exist and they are important components of immune regulation, their exact mechanisms of action have not yet been determined. There are five studies in the literature evaluating the status of soluble immune checkpoint molecules in breast cancer patients, with one being a review article. It is highly likely that immune checkpoint molecules found on both the cell surface and soluble in blood and body fluids are also present in tumor metastatic regions. There is no study using these immunological biomarkers to determine metastasis in invasive ductal carcinoma patients with metastatic axillary lymph nodes ın the literature. In this study, the investigators will evaluate the soluble levels of immune checkpoint molecules in washout fluids obtained from metastatic axillary lymph nodes and benign lymph nodes in patients with invasive ductal breast carcinoma, and will assess the effectiveness of these immune checkpoint molecules and the washout method in diagnosing metastasis.

DETAILED DESCRIPTION:
The most common cancer in women worldwide and the leading cause of death among those aged 20-59 is breast cancer. Invasive breast cancers are primarily classified as ductal and lobular. However, special types of invasive breast cancers, which constitute 10% of total cases, have been included in the current histological classification.

Invasive ductal carcinoma is the most frequently observed type among invasive breast cancers (80%) and is also defined as invasive ductal carcinoma of no special type. Macroscopic or microscopic axillary lymph node metastases have been detected in up to 25% of screening-diagnosed cases and up to 60% of symptomatic cases of invasive ductal carcinoma.

The clinical staging of breast cancer is primarily determined by the physical examination of the breast skin, breast tissue, and regional lymph nodes (axillary, supraclavicular, and internal mammary). However, the accuracy of clinically determining axillary lymph node metastases is only 33%. Proper lymph node staging in breast cancer patients is crucial for both prognosis and treatment.

Ultrasound is significantly more sensitive than physical examination alone in determining axillary lymph node involvement in breast cancer staging. For lymph nodes that remain indeterminate or suspicious on ultrasound, fine-needle aspiration biopsy or core biopsy provides a definitive diagnosis. The most commonly used staging system is the TNM staging system. The American Joint Committee on Cancer (AJCC) recently modified the TNM system. According to the latest TNM staging, the presence of macrometastases in ipsilateral level 1 and level 2 axillary lymph nodes classifies breast cancer as stage 2A or higher. Although biopsy sampling has a high diagnostic accuracy, it requires experienced pathologists, and the evaluation process can take weeks. Therefore, there is a need for faster and more cost-effective diagnostic methods for detecting axillary metastases.

The lymph node washout technique is used to determine lymph node metastasis in malignancies such as papillary thyroid carcinoma, the most common type of thyroid cancer. Papillary thyroid carcinomas generally do not exhibit aggressive clinical behavior and have favorable long-term prognoses. However, at the time of diagnosis, cervical and mediastinal lymph node involvement ranges from 27% to 46%, and the postoperative recurrence rate is between 3% and 30%. Thus, determining preoperative lymph node involvement and distinguishing it from benign reactive lymphadenitis is essential. For this purpose, fine-needle aspiration with thyroglobulin washout sampling has recently become widely used worldwide. In patients with papillary thyroid carcinoma, fine-needle aspiration of cervical lymph nodes and testing for thyroglobulin, a protein normally present in thyroid tissue, is considered one of the most reliable methods for detecting lymph node metastasis. A large-scale study by Moon et al. found that fine-needle aspiration thyroglobulin washout had a sensitivity of 93.2% and a specificity of 95.9% in detecting lymph node metastases in papillary thyroid carcinoma.

Immune checkpoints have gained attention, particularly after being awarded the Nobel Prize in 2018, as they play a crucial role in understanding the relationship between cancer and the immune system. PD-1 and its ligand PD-L1 function as immune checkpoints by inhibiting T-cell receptor signaling and co-stimulatory signals. T-cell immunoglobulin and mucin domain 3 (TIM-3) is expressed on interferon-γ-producing T cells, regulatory T cells (Tregs), dendritic cells, B cells, macrophages, natural killer (NK) cells, and mast cells. Dysregulation of TIM-3 expression has been linked to autoimmune diseases. High TIM-3 expression is associated with T-cell exhaustion and suppression of T-cell responses, particularly in chronic viral infections and tumor development. The clinical success of immune checkpoint inhibitors such as ipilimumab and nivolumab in melanoma and lung cancer has further increased interest in immune checkpoints.

Numerous studies in the literature have investigated the expression of immune checkpoints such as PD-1, PD-L1, and CTLA-4 on the cell surface in breast cancer patients. One study evaluating the genetic expression of immune checkpoints in breast cancer found a negative correlation between B7-H3 mRNA expression and survival, while a positive correlation was observed between survival and the expression of CTLA-4 and tyrosine-based inhibitory motif domain (TIGIT). Another study reported decreased Lymphocyte-activation gene 3 (LAG-3) expression in triple-negative breast cancer and human epidermal growth factor receptor 2 (HER2) positive breast cancers.

Natural soluble forms of immune checkpoint receptors and ligands also exist in body fluids and play a role in immune regulation, although their exact mechanisms remain unclear. Many studies are investigating the role of immune checkpoints in cancer patients. One study evaluated both tumor-associated and soluble levels of PD-L1 and CTLA-4 in the blood, finding that elevated levels of PD-L1 and CTLA-4 were associated with poor prognosis. There are five studies in the literature, including one report, evaluating soluble immune checkpoints in breast cancer patients.

Since immune checkpoints are present on the cell surface and in soluble form in blood and body fluids, they are also highly likely to be found in tumor-metastasized regions. In the literature there is no study using these immunological markers to determine metastasis in patients with invasive ductal carcinoma and metastatic axillary lymph nodes.

In this study, the investigators will evaluate the soluble levels of immune checkpoints commonly associated with cancer-sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active Transforming growth factor (TGF)-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, and Galectin-9-in washout fluid samples obtained from metastatic axillary lymph nodes and benign lymph nodes in patients with invasive ductal breast carcinoma. The effectiveness of immune checkpoints and the washout technique in diagnosing lymphatic metastasis will be assessed as a rapid diagnostic method.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven invasive ductal carcinoma
* Patients who will have neoadjuvant therapy

Exclusion Criteria:

* The fine-needle aspiration biopsy (FNAB) result of the suspected metastatic lymph node is negative.
* The FNAB result of the presumed healthy lymph node is malignant.
* They refuse to participate in the study.
* They have another primary malignancy.
* They are pregnant.
* They have a history of immunodeficiency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The immune checkpoints in lymph node washout fluid | 3 monthts
  The immune checkpoints (sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active Transforming growth factor (TGF)-β1, The cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), Programmed death ligand 1 (PD-L1), Programmed cell death protein 1 (PD-1), T-cell immunoglobulin and mucin domain 3 (Tim-3), Lymphocyte-activation gene 3 (LAG-3), and Galectin-9) will be measured at lymph node washout fluid and the results will be presented in pg/ml.

SECONDARY OUTCOMES:
The immune checkpoints in blood | 3 monthts
  The immune checkpoints (sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active Transforming growth factor (TGF)-β1, The cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), Programmed death ligand 1 (PD-L1), Programmed cell death protein 1 (PD-1), T-cell immunoglobulin and mucin domain 3 (Tim-3), Lymphocyte-activation gene 3 (LAG-3), and Galectin-9) will be measured at serum samples and the results will be presented in pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giuliano AE, Connolly JL, Edge SB, Mittendorf EA, Rugo HS, Solin LJ, Weaver DL, Winchester DJ, Hortobagyi GN. Breast Cancer-Major changes in the American Joint Committee on Cancer eighth edition cancer staging manual. CA Cancer J Clin. 2017 Jul 8;67(4):290-303. doi: 10.3322/caac.21393. Epub 2017 Mar 14. PMID 28294295
- [Background] Moon JH, Kim YI, Lim JA, Choi HS, Cho SW, Kim KW, Park HJ, Paeng JC, Park YJ, Yi KH, Park DJ, Kim SE, Chung JK. Thyroglobulin in washout fluid from lymph node fine-needle aspiration biopsy in papillary thyroid cancer: large-scale validation of the cutoff value to determine malignancy and evaluation of discrepant results. J Clin Endocrinol Metab. 2013 Mar;98(3):1061-8. doi: 10.1210/jc.2012-3291. Epub 2013 Feb 7. PMID 23393171
- [Background] Sallout L, Tashkandi M, Moqnas A, AlMajed H, Al-Naeem A, Alwelaie Y. Fine-needle aspiration biopsy of axillary lymph nodes: A reliable diagnostic tool for breast cancer staging. Cancer Cytopathol. 2024 Feb;132(2):103-108. doi: 10.1002/cncy.22770. Epub 2023 Oct 16. PMID 37843531